CLINICAL TRIAL: NCT06975943
Title: Comparison in Cervical Length and Prolongation of Gestation Age on Vaginal Progesterone Administration to Pregnant Women After the Acute Phase of Threatened Preterm Birth : A Randomised Clinical Trial
Brief Title: Comparison in Cervical Length and Prolongation of Gestation Age on Vaginal Progesterone Administration to Pregnant Women After the Acute Phase of Threatened Preterm Birth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0976/KEPK/V/2024
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnant Women; Pregnancies at Increased Risk of Preterm Birth
Keywords: Interventional; Pregnant Women; Preterm Birth; Vaginal Progesterone; Indonesia
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive standard tocolytic treatment, receiving oral nifedipine for 48 hours in conjunction with dexamethasone injections to promote fetal lung development. Participants will have no progesterone treatment following arrested preterm labor. Monitoring for compliance will be conducted throughout the study period.
- Vaginal Progesterone (Active Comparator): This group will receive standard tocolytic treatment, receiving oral nifedipine for 48 hours in conjunction with dexamethasone injections to promote fetal lung development. Participants will receive daily vaginal micronized progesterone (Microgest®) of dose 200 mg for a duration of two weeks following arrested preterm labor. Monitoring for compliance and potential side effects will be conducted throughout the study period.
  Interventions: Drug: Progesterone 200 mg vaginal capsules

INTERVENTIONS:
Drug: Progesterone 200 mg vaginal capsules — Participants in this group will receive daily vaginal micronized progesterone (Microgest®) of dose 200 mg for a duration of two weeks following arrested preterm labor. This micronized progesterone will be administered to assess its impact on pregnancy prolongation and changes of cervical length following arrested preterm labor.
  Other Names: Microgest
  Arms: Vaginal Progesterone

SUMMARY:
This randomised clinical trial aims to investigate the effect of daily vaginal progesterone supplementation on pregnancy prolongation and cervical length changes following arrested preterm labor in singleton pregnancies. The study will recruit pregnant women between 28 and 33 weeks of gestational age who had experienced threatened preterm labor at Dr. Soetomo Hospital in Indonesia. Participants will be randomly divided into two groups: a Treatment Group receiving vaginal progesterone therapy and a Control Group receiving standard care without progesterone intervention. The primary outcomes are the prolongation of gestational age until delivery and the changes in cervical length over time. The secondary outcomes are recurrence of threatened preterm labor, mode of delivery, neonatal outcomes, and survival analysis. This study will provide valuable evidence supporting the use of vaginal progesterone as an effective intervention for women at risk of preterm labor and potentially improving maternal and neonatal outcomes in Indonesia and globally. All participants will be provided with detailed information about the study, and their participation will be voluntary. Ethical considerations, including informed consent and data confidentiality, will be strictly adhered to throughout the study.

DETAILED DESCRIPTION:
This prospective, open-label, randomised clinical trial aims to investigate the effect of daily vaginal progesterone supplementation on pregnancy prolongation and cervical length changes following arrested preterm labor in singleton pregnancies. Threatened preterm labor is characterised by rhythmic uterine contractions occurring without substantial cervical changes, as assessed through digital pelvic examination. The gestational age will be verified via ultrasound metrics and review of antenatal care documentation. All subjects will receive standard tocolytic treatment, oral nifedipine for 48 hours in conjunction with dexamethasone injections to promote fetal lung development. The arrest of preterm labor is characterised by a stable condition that does not advance to active labor, specifically defined as two or fewer contractions per ten minutes, intact membranes, and cervical dilatation of three centimetres or less, following a minimum of 48 hours after the first dose of tocolytics. Women will be enrolled 48 hours after tocolytic initiation. Upon obtaining written informed consent from the participants, baseline data will be collected for each individual. The baseline data comprise demographic and clinical information, including risk factors, digital pelvic examinations, and ultrasound findings. All participants will receive a digital pelvic examination to assess cervical dilation and effacement, as well as a transvaginal ultrasound to measure cervical length. Cervical length will be assessed by Ernawati at Dr. Soetomo Hospital utilising a standard procedure with a probe encased in a disposable cover, which is then inserted vaginally with an empty bladder. The cervical length will be reassessed at outpatient clinic visits at 7 days and 14 days post-enrollment. Subsequent to the acquisition of baseline data, all participants will be randomly allocated into two groups: the Control Group, which does not receive therapy, and the Therapy Group, which will receive vaginal progesterone. Ethical considerations are of utmost importance in this study. The study protocol will undergo evaluation and approval by an Institutional Review Board (IRB) or equivalent ethical committee. Confidentiality of participants will be preserved during the study, and data will be anonymised throughout analysis and reporting. All potential hazards related to the examination or drug administration will be comprehensively communicated to participants, and suitable safety protocols will be established. Participants will be notified of their right to withdraw from the study at any period without penalty.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnant women who have passed the acute phase of Threatened Preterm Labor that meets the following criteria:

   1. Persistent contractions (2-3 contractions in 10 minutes) accompanied by cervical dilation assessed based on pelvic examination (Vaginal Touche)
   2. Intact amniotic membrane
   3. Cervical dilation ≤ 2 cm
   4. No birth occurs within 2x24 hours since persistent contractions appear.
2. Age 18-40 years
3. The gestational age must be between 28 weeks and 33 weeks plus 6 days.
4. Able to participate, communicate well with researchers, and willing to provide written consent to participate in the study.

Exclusion Criteria:

1. Patients with cervical cerclage in this pregnancy
2. Cervical length is less than 10 mm
3. Congenital abnormalities in the fetus
4. Anatomical abnormalities in the uterus
5. History of antepartum hemorrhage in this pregnancy
6. Known hypersensitivity to progesterone or contraindications to its use.
7. Suspected or proven premature rupture of membranes at enrollment
8. Subjects on drug therapy known to interact with progesterone (eg Bromocriptine, Rifampin, Ketoconazole, and Cyclosporine)
9. Subjects with comorbidities: cardiovascular disease, renal function, liver function, hematological disorders, and other uncontrolled comorbidities.
10. Subjects with stress conditions based on the DASS-42 questionnaire.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 48 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Prolongation of Gestation Age | Enrollment and Delivery
  This measurement will be confirmed through ultrasound parameters and review of antenatal care records for gestation age at enrollment. Then the next measurement will be at delivery. Prolongation of gestation age will be measured in days.
Changes of Cervical Length | Enrollment, 7th and 14th day after enrollment
  This measurement will be confirmed through transvaginal ultrasound parameters at enrollment. The next measurement will be at subsequent obstetric clinic visits. Changes in cervical length will be measured in millimeters.

SECONDARY OUTCOMES:
Recurrence of Threatening Preterm Labor | 7th, 14th day after enrollment, and Delivery
  This measures the incidence of threatening preterm labor recurrence throughout the study.
Delivery Method | Delivery
  Delivery method will be categorized as spontaneous vaginal delivery, operative vaginal delivery, and cesarean section.
APGAR Score | Delivery
  This measure is a newborn health assessment system that is carried out by checking five vital criteria at the 1st and 5th minute. There are 5 parts to an Apgar score. Each category is weighted evenly and assigned a 0, 1, or 2 value. The components are then added to give a score recorded 1 and 5 minutes after birth. A score of 7 to 10 is considered reassuring, a score of 4 to 6 is moderately abnormal, and a score of 0 to 3 is deemed low in full-term and late preterm infants.
Baby Birth Weight | Delivery
  This measures the weight of the baby birth. The weight will be measured in grams.
NICU Admission | Delivery
  This measures how many newborns that was given intensive care.
Neonatal Mortality | Delivery and 28 days post partum
  This measures the number of fetal and newborn deaths under 28 days of age.

CONTACTS AND LOCATIONS:
Overall Officials: Ernawati Ernawati, Dr., Principal Investigator — Dr. Soetomo General Hospital Surabaya
Locations (1):
- Dr. Soetomo General Hospital Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
At this point, we remain undecided about disseminating Individual Participant Data (IPD) from this study to other researchers. Multiple elements are now being evaluated, encompassing the prospective advantages of data sharing for the enhancement of scientific knowledge, alongside the ethical and logistical problems related to safeguarding participant privacy and data security. We are assessing the criteria and regulations of prospective data repositories and funding organizations. A conclusive decision will be reached following thorough consideration and consultation with pertinent parties, including the Institutional Review Board (IRB) or ethical committee, and will be properly documented.